CLINICAL TRIAL: NCT02544282
Title: Large-scale Prospective Double-blind Randomized Controlled Trial of Pecs II Block for Breast Surgery: Effect on Postoperative Pain and Opioid Consumption
Brief Title: Large-scale Prospective Double-blind Randomized Controlled Trial of Pecs II Block for Breast Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GZA Ziekenhuizen Campus Sint-Augustinus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GZA-ANE-PECS-01
Record Dates: First submitted 2015-09-02; First posted 2015-09-09 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2015-10

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting
Keywords: Analgesics; Opioid; Mastectomy; Segmental Mastectomy; Pecs II
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Levobupivacaine; Sodium Chloride; Saline Solution; Sevoflurane; Propofol; Sufentanil; Atracurium; Acetaminophen; Tramadol; Pirinitramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pecs II (Active Comparator): General anesthesia followed by a Pecs II block and opioids if required
  Interventions: Drug: Levobupivacaine; Drug: Sevoflurane; Drug: Propofol; Drug: Sufentanil; Drug: Atracurium; Drug: Paracetamol; Drug: Tramadol; Drug: Piritramide
- Placebo (Placebo Comparator): General anesthesia followed by a placebo Pecs II block and opioids if required
  Interventions: Drug: NaCl 0.9%; Drug: Sevoflurane; Drug: Propofol; Drug: Sufentanil; Drug: Atracurium; Drug: Paracetamol; Drug: Tramadol; Drug: Piritramide

INTERVENTIONS:
Drug: Levobupivacaine — Pecs II Block
  Other Names: Chirocaine
  Arms: Pecs II
Drug: NaCl 0.9% — Placebo Pecs II block
  Other Names: Normal Saline
  Arms: Placebo
Drug: Sevoflurane — General Anesthesia
Drug: Propofol — General Anesthesia
Drug: Sufentanil — General Anesthesia
Drug: Atracurium — General Anesthesia
Drug: Paracetamol — Pain Relief
  Other Names: Acetaminophen
Drug: Tramadol — Pain Relief
Drug: Piritramide — Pain Relief

SUMMARY:
In this prospective trial, Stage 1-3 patients having mastectomies or isolated lumpectomy with axillary node dissection will be randomly assigned to general anesthesia with opioids combined with a Pecs II block or to general anesthesia with opioids combined with a placebo Pecs II block. Participants will be followed postoperatively during their entire hospital stay to determine the effectiveness of Pecs II block and opioids versus placebo Pecs II block and opioids as postoperative pain treatment.

DETAILED DESCRIPTION:
Each year, 9400 new cases of breast cancer are diagnosed in Belgium. It makes breast cancer the most common cancer in women, good for more than one third of all cancer cases in women.

Surgical excision of the tumour is a necessary and effective step to cure from the disease. Recent studies have demonstrated the positive effects of regional anesthesia on peroperative and postoperative pain. Paravertebral blocks have become popular as an alternative to the analgesia provided by the 'gold standard' of thoracic epidural analgesia. However, both regional techniques have complications and slow learning curves that make them unsuitable for the large proportion of breast surgery patients who are treated on a day-stay basis. Recently, Rafael Blanco introduced the Pecs and Pecs II blocks, a practical alternative to both paravertebral and epidural blockade in the management of pain after breast surgery.

The investigators introduced the Pecs II block in their clinical practice. This study compares general anesthesia with a Pecs II block to general anesthesia with a placebo Pecs II block for breast surgery. The objective is to evaluate analgesic effectiveness and changes in opioid consumption when applying a Pecs II block versus a placebo Pecs II block.

Stage 1-3 patients having mastectomies or tumourectomies with axillary clearance will be randomly assigned to general anesthesia with a Pecs II block or to general anesthesia with a placebo Pecs II block. Enrolling 140 patients over an anticipated time frame of 2 years will provide an 90% power and a p-value of 0.05 for perioperative and postoperative opioid consumption as well as pain scores (NRS). Confirming the hypothesis will indicate that a minor modification to the anesthetic procedure will reduce the opioid consumption (including it's unwanted side effects) during and after surgery while maintaining or reducing patients' indicated pain scores (NRS).

ELIGIBILITY:
Inclusion Criteria:

* Primary breast cancer without known extension beyond the breast and axillary nodes (i.e. believed to be Tumor Stage 1-3, Nodes 0-2)
* Scheduled for unilateral or bilateral mastectomy with or without implant (isolated "lumpectomy" will not qualify)
* Isolated "lumpectomy" with axillary node dissection (anticipated removal of at least five nodes)
* Written informed consent, including willingness to be randomized to opioids or regional analgesia
* Dutch speaking

Exclusion Criteria:

* Previous surgery for breast cancer (except diagnostic biopsies)
* Inflammatory breast cancer
* Scheduled free flap reconstruction
* ASA Physical Status ≥ 4
* Any contraindication to locoregional analgesia (including coagulopathy, abnormal anatomy)
* Any contraindication to midazolam, propofol, sevoflurane, sufentanyl, tramadol or piritramide
* Other cancer not believed by the attending surgeon to be in long-term remission
* Systemic disease believed by the attending surgeon to present ≥ 25% two-year mortality
* Obesity defined as BMI ≥ 30 kg/m2
* Chronic use of pain medication (started > 3 months ago)
* Allergic to Chirocaine
* Chronic drug or alcohol abuse
* INR > 1.4
* Thrombocytopenia < 70,000 platelets
* Dementia
* Pregnancy
* Kidney or liver failure

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | up to 72 hours after completion of surgery
  Within first hour: Each ten minutes by Recovery Nurse. Hour 2 till discharge ( max 72 hours post surgery): hourly by patient through questionnaire.Master data set is administrated by secretarial office of Anesthesia departement

SECONDARY OUTCOMES:
Peroperative Opioid Consumption | Peroperative period (max. 5 hours)
  Anesthetist in charge reports Opioid Consumption. Master data set is administrated by secretarial office of Anesthesia department
Postoperative Opioid Consumption | up to 72 hours after completion of surgery
  Nurse of postoperative recovery room and nurse of ward in charge reports opioid consumption on patient questionnaire. Master data set is administrated by secretarial office of Anesthesia department
Postoperative Nausea and Vomiting | up to 72 hours after completion of surgery
  Nurse of postoperative recovery room and nurse of ward in charge reports patients nausea and vomiting as well as the administered medication against postoperative nausea and vomiting on patient questionnaire. Master data set is administrated by secretarial office of Anesthesia department

CONTACTS AND LOCATIONS:
Overall Officials: Barbara JB Versyck, MD, Principal Investigator — GZA Ziekenhuizen Campus Sint-Augustinus
Locations (1):
- GZA Sint Augustinus, Wilrijk, Antwerpen, Belgium

REFERENCES:
- [Result] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099